CLINICAL TRIAL: NCT05611606
Title: Welfare Benefits for Individuals With Functional Somatic Disorders: DanFunD
Brief Title: Welfare Benefits in Functional Somatic Disorders
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Center for Clinical Research and Prevention (Network)
Responsible Party: Sponsor
Other Study IDs: DanFunD welfare benefits
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-10

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Chronic Fatigue Syndrome; Bodily Distress Syndrome; Somatoform Disorders; Medically Unexplained Syndrome; Medically Unexplained Symptoms
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Fatigue Syndrome, Chronic; Somatoform Disorders; Medically Unexplained Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DanFunD baseline: Data from the DanFunD baseline cohort will be included (11). It comprises a total of 9,656 (33.7% of the invited participants) men and women aged 18-76 years born in Denmark and living in the Western part of greater Copenhagen.
  Individuals with FSD are identified by means of self-reported questionnaires (n=9,656) (2) and diagnostic research interviews (n=1,590) (12).
  Participants with FSD will be defined as follows:
  * FSD operationalised by the Bodily Distress Syndrome single- and multi-organ type will be defined with both self-reported questionnaires (14) and diagnostic interviews (3)
  * Three functional somatic syndromes, i.e. irritable bowel (15), chronic widespread pain (16), and chronic fatigue (17) will be defined with questionnaires.
  Severe physical disease will be defined as having received at least one of the following five diagnoses: Cancer, stroke, myocardial infarction, other heart disease, and obstructive pulmonary disease.

SUMMARY:
The objective of this observational study is to estimate the number of weeks of welfare benefits, i.e. sickness benefit, unemployment benefit and social assistance, for individuals with functional somatic disorders and compare them to

1. healthy individuals, and
2. individuals with severe physical disease.

DETAILED DESCRIPTION:
Functional somatic disorders (FSD) are common conditions characterized by persistent patterns of physical symptoms that cannot be better explained by other physical or mental conditions (1). The conditions may cause severe impairment for the patients who present with reduced physical and mental health, lower social status, and poor labour market association (2-4).

In 2005, it was estimated that FSD accounted for 3% of hospitalizations and 10-20% of health care expenses in Denmark (5), and a newer Danish primary care study has shown patients with FSD to have higher annual health care costs compared with conventionally-defined conditions (6). In other countries, studies in clinical samples have shown increased direct and indirect health care costs of FSD (7, 8) showing a dose-response relationship with severity of the FSD (9). These studies into highly selected clinical samples may induce high risk of selection bias, and studies including random selected general population samples are therefore needed. One Canadian population-based study on health care costs of children, adolescents, and young adults with FSD also found increased health care use and costs for this group (10). Studies investigating the socioeconomic burden in terms of welfare benefits of FSD in an adult random sample from the general population are, however, lacking.

Objective To estimate the number of weeks of welfare benefits, i.e. sickness benefit, unemployment benefit and social assistance, for individuals with FSD and compare them to individuals without FSD and individuals with severe physical disease.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* Not born in Denmark
* Not being a Danish citizen
* Pregnancy

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were randomly drawn from the adult general Danish population by means of the the Danish Civil Registration system.
  The DanFunD baseline cohort comprises a total of 9,656 (33.7% of invited participants) men and women aged 18-76 years, born in Denmark, and living in the Western part of greater Copenhagen. All participants filled in questionnaires regarding physical symptoms and psychological factors, among others. A stratified subsample (n=2,450) of every tenth participant and every symptom high score participant on the DanFunD baseline symptom questionnaires were invited to participate in a diagnostic interview, the Research Interview for Functional somatic Disorders (RIFD), performed by trained family physicians (28); 1,590 (64.9%) accepted and participated in the interview.
Sampling Method: Probability Sample
Enrollment: 9656 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Sickness benefit | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  Wellfare benefit disbursed to employed citizens being ill, unemployed citizens currently ill, citizens in activation programs currently ill, and citizens in flexible jobs but currently ill
Unemployment benefit | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  Welfare benefit disbursed to unemployed citizens who receive unemployment benefit (full or part time, during vacation or activation) together with citizens on social assistance who are deemed ready-to-work, only receiving social assistance because of unemployment, but having no entitlement to unemployment benefit.
Social assistance | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  A welfare payment administered by the municipal social service department and is allocated if citizens are unable to support themselves.

SECONDARY OUTCOMES:
No transfer income/self-support | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  Individuals that do not receive welfare payments under the circumstances of sickness, unemployment, or social benefits. Including leave-of-absence schemes and grants from State Education Fund.
Public retirement pension | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  Public retirement pension
Emigration | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  Participant not resident in Denmark
Death | 10-year period before and 5-year period after the day the participant participated in the DanFunD baseline investigation
  Participant dead

CONTACTS AND LOCATIONS:
Overall Officials: Per Fink, DMSc, Study Chair — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petersen MW, Wellnitz KB, Carstensen TBW, Dantoft TM, Ornbol E, Bjerregaard AA, Jorgensen T, Fink P. Welfare benefit utilization for people with functional somatic disorder. A population-based cohort study. J Psychosom Res. 2025 Apr;191:112073. doi: 10.1016/j.jpsychores.2025.112073. Epub 2025 Feb 27. PMID 40037070

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT05611606/SAP_000.pdf